CLINICAL TRIAL: NCT03776747
Title: Repeatability in Hyperpolarized 3-Helium Magnetic Resonance Imaging
Brief Title: Repeatability in Hyperpolarized 3-Helium With MRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eric A. Hoffman (Other)
Responsible Party: Sponsor-Investigator, Eric A. Hoffman, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200803776
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Radiation Exposure
MeSH Terms: interventions — Contrast Media; Respiratory Function Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group One: Prone MRI Scans (Experimental): Subjects will have vitals, pulmonary function tests, initial proton MRI scan, prone hyperpolarized 3 helium gas scan
  Interventions: Drug: Prone hyperpolarized 3 helium gas scan; Diagnostic Test: Vitals; Diagnostic Test: Pulmonary Function Tests; Diagnostic Test: Initial protocol MRI scan
- Group Two: Supine MRI scans (Active Comparator): Subjects will have vitals, pulmonary function tests, initial protocol MRI scan, supine hyperpolarized 3 helium gas scan
  Interventions: Drug: Supine hyperpolarized 3 helium gas scan; Diagnostic Test: Vitals; Diagnostic Test: Pulmonary Function Tests; Diagnostic Test: Initial protocol MRI scan

INTERVENTIONS:
Drug: Prone hyperpolarized 3 helium gas scan — Hyperpolarized gas used as a contrast agent to test reproducibility of MRI of the lungs/Images done while subject is prone.
  Other Names: Prone MRI scan with contrast
  Arms: Group One: Prone MRI Scans
Drug: Supine hyperpolarized 3 helium gas scan — Hyperpolarized gas used as a contrast agent to test reproducibility of MRI of the lungs/Images done while subject is supine.
  Other Names: Supine MRI scan with contrast
  Arms: Group Two: Supine MRI scans
Diagnostic Test: Vitals
Diagnostic Test: Pulmonary Function Tests — Pre and post spirometry, diffuse lung carbon monoxide (DLCO), lung volumes
Diagnostic Test: Initial protocol MRI scan — Initial scan to determine placement

SUMMARY:
The main purpose of this study is to assess and test the reproducibility and results of hyperpolarized 3-Helium gas as a contrast agent with Magnetic Resonance Imaging (MRI) of the lungs in healthy adult subjects.

DETAILED DESCRIPTION:
New CT imaging techniques often expose the patient to higher doses of radiation. There is a great deal of concern about effects of medical radiation exposure on the general public and regulations are becoming stricter on the radiation doses that are allowed.

One novel procedure that has been developed to evaluate the function and structure of the lung is the use of hyperpolarized gases with MRI scanners. We want to compare the lung imaging techniques that we have developed in our lab to a technique that uses hyperpolarized 3-Helium gas with MRI. This technique is free from radiation and less invasive than many lung imaging techniques.

Hyperpolarized gas MRI is based on the introduction of spins into the lungs, allowing imaging to take place. The use of hyperpolarized 3-Helium has a few advantages:

1. it allows us to see the microstructure of the lungs through diffusion imaging (apparent diffusion coefficient) which correlates with the size of airways and alveolar space.
2. it allows us to see ventilation, or how air moves in the lungs, at a high resolution.
3. it is capable of ultra fast imaging which will help us assess gas flow patterns within the airways.

and 4) the speed of depolarization lets us measure the partial pressure of oxygen and associated gas exchange mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* must be between the ages of 18 and 90
* must have a Body Mass Index (BMI) of < 32 and weigh < 200 lbs.

Exclusion Criteria:

* if female, must not be pregnant or breastfeeding
* must not have any metal objects in or on their body including body piercings that cannot be easily removed, bullets, metallic fragments or slivers in eyes, skin, etc., pacemaker or defibrillation, aneurysm clips, cochlear implants, coronary stents, or neurostimulation.
* must not have a history of claustrophobia, panic disorders, anxiety attacks, atrial fibrillation, uncontrolled high blood pressure, frequent ventricular ectopic rhythm, hemodynamic instability, kidney dysfunction or heart disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-07-22 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Hoffman, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group One: Prone MRI Scans: Subjects will have vitals, pulmonary function tests, initial proton MRI scan, prone hyperpolarized 3 helium gas scan
  Prone hyperpolarized 3 helium gas scan: Hyperpolarized gas used as a contrast agent to test reproducibility of MRI of the lungs/Images done while subject is prone.
  Vitals
  Pulmonary Function Tests: Pre and post spirometry, diffuse lung carbon monoxide (DLCO), lung volumes
  Initial protocol MRI scan: Initial scan to determine placement
- Group Two: Supine MRI Scans: Subjects will have vitals, pulmonary function tests, initial protocol MRI scan, supine hyperpolarized 3 helium gas scan
  Supine hyperpolarized 3 helium gas scan: Hyperpolarized gas used as a contrast agent to test reproducibility of MRI of the lungs/Images done while subject is supine.
  Vitals
  Pulmonary Function Tests: Pre and post spirometry, diffuse lung carbon monoxide (DLCO), lung volumes
  Initial protocol MRI scan: Initial scan to determine placement
Period: Overall Study
Arm/Group | Group One: Prone MRI Scans | Group Two: Supine MRI Scans
Started | 0 | 18
Completed | 0 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only supine MRI subjects were recruited
Groups:
- Total: Total of all reporting groups
Arm/Group | Group One: Prone MRI Scans | Group Two: Supine MRI Scans | Total
Number analyzed (Participants) | 0 | 18 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 17 | 17
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 8 | 8
  Male |  | 10 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States |  | 18 | 18

OUTCOME MEASURES:

1. Primary Outcome: Apparent Diffusion Coefficient (ADC) as a Function of Lung Inflation Levels.
Description: Validate the intrinsic variability of ADC (cm2/s) as a function of normal procedural and physiological changes in an attempt to standardize the use of the biomarker in future assessments of pulmonary pathologies.
Time Frame: Through study completion, measurements completed at one day visit only.
Population: Only Supine MRI's were performed. ADC values at 20%, 60% and 100% vital capacity (VC) were compared against each other.
Measure: Mean (Standard Deviation); unit: ADC (cm2/sec)
Arm/Group | Group One: Prone MRI Scans | Group Two: Supine MRI Scans
Number analyzed (Participants) | 0 | 18
ADC (cm2/sec)
  20% VC |  | 0.167 (.018)
  60% VC |  | 0.175 (.015)
  100% VC |  | 0.188 (.020)
Statistical Analysis 1: Comparison: Group Two: Supine MRI Scans; We hypothesized that the anisotropic deformation index (ADC) is dependent upon lung inflation level. (Thus, it is important to standardize lung inflation when using this method); Test type: Other — Analysis of variance between lung inflation levels; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 weeks.
Description: There were no adverse events reported.
Arm/Group | Group One: Prone MRI Scans | Group Two: Supine MRI Scans
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/18
Other Adverse Events (participants affected / at risk) | 0/0 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No